CLINICAL TRIAL: NCT06485960
Title: Validation of the Experience Sampling Dietary Assessment Method (ESDAM)
Brief Title: Validation of the Experience Sampling Dietary Assessment Method
Acronym: YONAS
Status: Recruiting | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Christophe Matthys, Professor dr., KU Leuven
Other Study IDs: S68363; C3/22/050 (Other Grant/Funding Number: KU Leuven)
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-08

CONDITIONS: Validation Study
Keywords: Dietary assessment; Validation; Experience Sampling; digital health; digital biomarkers; doubly-labeled water; ESM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- YONAS 1: ESDAM validation
  Interventions: Other: ESDAM validation

INTERVENTIONS:
Other: ESDAM validation — * 3* 24-Hour Dietary Recalls
  * Experience Sampling Dietary Assessment Method (mobile application)
  * Continuous Blood Glucose Monitoring
  * Wrist- worn motion sensors
  * Doubly-labeled water administration
  * Blood drawings (Erythrocyte Membrane Fatty Acid composition, Carotenoids, polyphenols)
  * Urine sampling (Doubly-labeled water, urinary nitrogen)

SUMMARY:
A new dietary assessment method was developed based on the Experience Sampling Methodology. In order to use this newly developed Experience Sampling Dietary Assessment Method (ESDAM) in research and clinical practice as a valid and reliable method to measure dietary intake the ESDAM needs to be validated against objective biomarkers and reference methods.

DETAILED DESCRIPTION:
The purpose of this research project is to advance nutritional research by delivering an improved, accurate, feasible and reliable method to assess dietary intake. Our newly developed approach to collate dietary intake based on experience sampling methodology (ESM) will serve this purpose.

Therefore, this research aims to validate the newly developed Experience Sampling Dietary Assessment Method (ESDAM) by assessing construct validity compared to blood and urine biomarkers representing dietary intake. This will eventually result in the newly developed dietary assessment method being evidence-based and validated and, thus, ready-to-use as a reliable method for research and clinical practice.

Therefore, the ESDAM will be validated against repeated 24-hour dietary recalls, the doubly-labelled water method, urinary nitrogen and blood biomarkers. The study has a duration of four weeks. The first two weeks will be used to collect baseline data including socio-demographic, biometric data and three 24-hour recalls to assess dietary intake. During the last two weeks the Experience Sampling Dietary Assessment Method will be evaluated against urine biomarkers (Doubly-labeled water and urinary nitrogen), blood biomarkers (erythrocyte membrane fatty acid composition, beta-carotenoids, polyphenols) together with continuous glucose monitoring and two wrist-worn motion sensor devices to track eating- related movements.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Having a smartphone and being capable of using the smartphone and apps
* Having a freezer at home
* Sufficient knowledge of the Dutch language to understand and participate in the study
* Having a stable body weight (body weight not changed by 5% last 3 months)
* Not aiming to gain or lose weight during the study period

Exclusion Criteria:

* Pregnant or lactating women
* Not following a specific diet for medical reasons (i.e. coeliac disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Daily dietary energy intake based on the Experience Sampling Dietary Assessment Method | 2 weeks
  Daily dietary energy intake estimated by the Experience Sampling Dietary Assessment Method (ESDAM) compared to the Doubly-labeled Water Method
Daily dietary protein intake based on the Experience Sampling Dietary Assessment Method | 2 weeks
  Daily dietary protein intake estimated by the Experience Sampling Dietary Assessment Method (ESDAM) compared to urinary nitrogen
Daily energy expenditure derived from the doubly-labeled water method | 2 weeks
  Daily energy expenditure (kcal/day) measured by the doubly-labeled water method
Daily dietary protein intake based on urinary nitrogen analysis | 2 weeks
  Daily dietary protein intake based on urinary nitrogen analysis

SECONDARY OUTCOMES:
Dietary intake based on Experience Sampling Dietary Assessment Method | 2 weeks
  Daily nutrient and food group consumption estimated by the Experience Sampling Dietary Assessment Method ESDAM
Dietary intake based on 24-hour dietary recalls | 2 weeks
  Energy, nutrient and food group consumption measured by the 24-hour dietary recalls
Serum Beta-carotenoid concentration | 4 weeks
  Serum Beta-carotenoids as biomarker of fruit and vegetable consumption
Erythrocyte membrane fatty acid composition | 4 weeks
  Erythrocyte membrane fatty acid composition as biomarker of fatty acid consumption
Plasma polyphenol concentration | 4 weeks
  Plasma polyphenol concentration as an indication of dietary polyohenol intake

OTHER OUTCOMES:
Timing of glucose peaks | 2 weeks
  Timing of glucose peaks registered by Continuous Glucose Monitoring
Timing of eating-related motion | 2 weeks
  Timing of eating-related motion monitored by wrist-worn motion sensors

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Matthys, PhD, Principal Investigator — KU Leuven/UZ Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verbeke J, Verbeke K, Van der Schueren B, Vangoitsenhoven R, Matthys C. Protocol of the validation of the experience sampling-based dietary assessment method (ESDAM) against doubly labeled water, urinary protein, and biomarkers. Nutr J. 2025 Nov 5;24(1):169. doi: 10.1186/s12937-025-01232-3. PMID 41194100